CLINICAL TRIAL: NCT00810225
Title: CNDP1 Polymorphisms in Gulf War Illness (GWI)
Brief Title: Study of Gulf War Illness (GWI) by Comparing GWI and Healthy Veterans
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Baraniuk, MD, Professor of Medicine, Georgetown University
Other Study IDs: 2008-012; USAMRMC PR# W81XWH-07-1-0618; HRPO Log No. A-14542.1
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Gulf War Illness; Persian Gulf War Syndrome
Keywords: CNDP1; carnosine dipeptidase 1; Persian Gulf War; Gulf War Syndrome; GWI; Gulf War Illness; Exercise; Chronic Fatigue; Fibromyalgia; Veterans; Irritable Bowel Syndrome; Migraine headaches; Neuropathy; Multiple Chemical Sensitivity
MeSH Terms: conditions — Persian Gulf Syndrome; Motor Activity; Fibromyalgia; Irritable Bowel Syndrome; Migraine Disorders; Multiple Chemical Sensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, and buccal swab samples retained for testing as described in protocol.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: GWI: veterans of the 1990-1991 Persian Gulf War who have autonomic, neurological and other symptoms
- 2: HC: healthy veterans of the 1990-1991 Persian Gulf War

SUMMARY:
Determine if:

* genetic differences of CNDP1 gene
* the previously defined GWI/Chronic Fatigue Syndrome (GWI/CFS) cerebrospinal fluid proteome contents
* psychometric
* other variables can differentiate between veterans of the 1990-1991 Persian Gulf War who have autonomic, neurological and other symptoms and those without these complaints.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of military enlistment between August 1, 1990 and July 31, 1991, and deployment for 30 consecutive days to:

  * Persian Gulf waters and adjacent land areas
  * Other global locations
  * U.S. only
* Status prior to 1990 and 1991:

  * Active duty
  * National Guard
  * Reserves

Exclusion Criteria:

* Current active duty military personnel
* Any one who was not active duty military personnel between August 1, 1990 and July 31, 1991
* HIV/AIDS; pregnancy or lactation; potential hepatitis; drug addiction; chronic inflammatory, infectious, or autoimmune medical illnesses not associated with GWI; incarceration; dementia, other cognitive limitation; or reliance on a care-giver in order to respond to the questionnaires and other study tests.

Amputations of one or both hands and forearms will be permitted but hand grip tests will not be tested

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All veterans who served in the Armed Forces between August 1990 and July 1991
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Baraniuk, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Gray GC, Reed RJ, Kaiser KS, Smith TC, Gastanaga VM. Self-reported symptoms and medical conditions among 11,868 Gulf War-era veterans: the Seabee Health Study. Am J Epidemiol. 2002 Jun 1;155(11):1033-44. doi: 10.1093/aje/155.11.1033. PMID 12034582
- [Background] Baraniuk JN, Casado B, Maibach H, Clauw DJ, Pannell LK, Hess S S. A Chronic Fatigue Syndrome - related proteome in human cerebrospinal fluid. BMC Neurol. 2005 Dec 1;5:22. doi: 10.1186/1471-2377-5-22. PMID 16321154
- [Background] Janssen B, Hohenadel D, Brinkkoetter P, Peters V, Rind N, Fischer C, Rychlik I, Cerna M, Romzova M, de Heer E, Baelde H, Bakker SJ, Zirie M, Rondeau E, Mathieson P, Saleem MA, Meyer J, Koppel H, Sauerhoefer S, Bartram CR, Nawroth P, Hammes HP, Yard BA, Zschocke J, van der Woude FJ. Carnosine as a protective factor in diabetic nephropathy: association with a leucine repeat of the carnosinase gene CNDP1. Diabetes. 2005 Aug;54(8):2320-7. doi: 10.2337/diabetes.54.8.2320. PMID 16046297
- [Background] Casado B, Zanone C, Annovazzi L, Iadarola P, Whalen G, Baraniuk JN. Urinary electrophoretic profiles from chronic fatigue syndrome and chronic fatigue syndrome/fibromyalgia patients: a pilot study for achieving their normalization. J Chromatogr B Analyt Technol Biomed Life Sci. 2005 Jan 5;814(1):43-51. doi: 10.1016/j.jchromb.2004.09.056. PMID 15607706
- [Background] Fukuda K, Nisenbaum R, Stewart G, Thompson WW, Robin L, Washko RM, Noah DL, Barrett DH, Randall B, Herwaldt BL, Mawle AC, Reeves WC. Chronic multisymptom illness affecting Air Force veterans of the Gulf War. JAMA. 1998 Sep 16;280(11):981-8. doi: 10.1001/jama.280.11.981. PMID 9749480
- [Derived] Narayan V, Shivapurkar N, Baraniuk JN. Informatics Inference of Exercise-Induced Modulation of Brain Pathways Based on Cerebrospinal Fluid Micro-RNAs in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. Netw Syst Med. 2020 Nov 18;3(1):142-158. doi: 10.1089/nsm.2019.0009. eCollection 2020. PMID 33274349
- See also: Laboratory Website — http://www9.georgetown.edu/faculty/baraniuj/Site/Welcome.html